CLINICAL TRIAL: NCT04649450
Title: MusiC to Prevent deliriUm During neuroSurgerY: A Single Centered Prospective Randomized Controlled Trial
Brief Title: MusiC to Prevent deliriUm During neuroSurgerY
Acronym: MUSYC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, A.J.P.E. VIncent, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2020-0064
Record Dates: First submitted 2020-09-11; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Delirium
Keywords: Neurosurgery; Delirium; Music; Randomized Controlled Trial
MeSH Terms: conditions — Delirium | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to either the intervention (music) or control (standard care) group.
Masking Description: Music vs. standard clinical care. No blinding of treatment was conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Participants in the music group will receive headphones with music 30 minutes before surgery. Patients will be able to choose music from a preselected list composed by a team consisting of researchers and dedicated music therapists. The headphones will be removed before entering the operating room. Once in the operating room they will receive earphones after intubation, compatible with the Mayfield and site of operation. The intraoperative music intervention will be continued during the surgical procedure and discontinued just before detubation. The duration of the intraoperative music intervention depends on the duration of surgery and will be documented. After surgery, during recovery at the post-operative care unit (PACU) another 30 minutes of music through headphones will be given. The following 3 days (post-operative day 1, 2 and 3) at the neurosurgical ward they will receive music twice a day for 30 minutes. All participants will further receive standard of clinical care.
  Interventions: Other: Music
- Standard of clinical care (No Intervention): Standard of clinical care.

INTERVENTIONS:
Other: Music — Participants in the music group will receive headphones with music 30 minutes before surgery. Patients will be able to choose music from a preselected list composed by a team consisting of researchers and dedicated music therapists. The headphones will be removed just before entering the operating room. Once in the operating room they will receive earphones after intubation, compatible with the Mayfield and site of operation. The intraoperative music intervention will be continued during the surgical procedure and discontinued just before detubation. The duration of the intraoperative music intervention depends on the duration of surgery and will be documented. After surgery, during recovery at the post-operative care unit (PACU) another 30 minutes of music through headphones will be given. The following 3 days at the neurosurgical ward they will receive music twice a day for 30 minutes.
  Arms: Music

SUMMARY:
Rationale: Delirium is a common and severe complication after neurosurgical procedures. Music before, during and after surgical procedures has proven its effectiveness in reducing pain, anxiety, stress and opioid medication in surgical patients. These symptoms belong to the main eliciting factors for developing delirium. Effective preventive therapy for delirium is not available. The investigators hypothesize that music listening, being a sustainable intervention with negligible risk of side effects, can lower delirium incidence among neurosurgical patients, resulting in reduction of in-hospital stays, healthcare costs and post-operative morbidity and mortality.

Objective: To assess the effect of peri-operative music on post-operative delirium in patients undergoing a craniotomy.

Study design: Single-centre prospective randomized controlled trial.

Study population: Adult patients undergoing a craniotomy at the Erasmus MC in Rotterdam.

Intervention: Recorded music, with headphones or earphones, before, during and after surgery.

Main study parameters/endpoints: Diagnosis of post-operative delirium screened by the DOS score confirmed by the consultant psychiatrist following the DSM-V criteria.

DETAILED DESCRIPTION:
Rationale:

Delirium is a common and severe complication after neurosurgical procedures. Music before, during and after surgical procedures has proven its effectiveness in reducing pain, anxiety, stress and opioid medication in surgical patients. These symptoms belong to the main eliciting factors for developing delirium. Effective preventive therapy for delirium is not available. The investigators hypothesize that music listening, being a sustainable intervention with negligible risk of side effects, can lower delirium incidence among neurosurgical patients, resulting in reduction of in-hospital stays, healthcare costs and post-operative morbidity and mortality.

Objective:

To assess the effect of peri-operative music on post-operative delirium in patients undergoing a craniotomy.

Hypothesis effect and sample size:

The investigators expect an incidence of delirium in our control group of 30%. This is based on literature documenting incidence of delirium in neurosurgical patients in a northern European population of 29-33%.The expected effect cannot be based on previous literature since no adequate trials exist on the effect of music on delirium. Other non-pharmacological interventions in delirium prevention mention a relative reduction of 36-77%. The investigators will consider the intervention clinical relevant if a relative reduction of 60% with an absolute reduction of 18% is achieved. Taking into account the incidence of delirium of 30%, a power of 80%, a two-sided significant p-value of <0,05 in a 1:1 randomization leads to a sample size of 90 patients per arm. The investigators expect a loss to follow-up of 5% and will therefore include 189 patients.

Interventions:

Patients will be randomly allocated to either the intervention (music) or control (standard care) group. Participants in the music group will receive headphones with music 30 minutes before surgery. Patients will be able to choose music from a preselected list composed by a team consisting of researchers and dedicated music therapists. The headphones will be removed just before entering the operating room. Once in the operating room they will receive earphones after intubation, compatible with the Mayfield and site of operation. The intraoperative music intervention will be continued during the surgical procedure and discontinued just before detubation. The duration of the intraoperative music intervention depends on the duration of surgery and will be documented. After surgery, during recovery at the post-operative care unit (PACU) another 30 minutes of music through headphones will be given. The following 3 days at the neurosurgical ward they will receive music twice per day for 30 minutes.

Primary outcome: The primary outcome measure is presence or absence of postoperative delirium within the first 5 days after surgery. All participating patients on the ward will be screened using the Delirium Observation Screening (DOS) scale. Additional to the DOS, in case of raised suspicion of delirium, a psychiatrist is consulted to confirm or reject clinical diagnosis of delirium based on the DSM-V criteria.

Secondary outcome:

* Severity and duration of delirium (DRS-R-98)
* Pre-operative anxiety (VAS-A)
* Activation of the parasympathetic nervous system measured with HRV.
* Depth of anaesthesia registered with Bispectral Index (BIS).
* Peri-operative medication use.
* Postoperative pain (NRS).
* Patients with postoperative complications (AE/SAE's).
* Hospital length of stay (days).
* Cognitive function (MoCA).
* Patient functional outcome (KPS).
* Patient functional outcome (mRS).
* Mortality and readmission rate.
* Patient-reported outcome (EORTC-QLQ-C30)
* Patient-reported outcome (EORTC-QLQ-BN20)
* Patient-reported outcome (EQ-5D).
* Patient satisfaction (VAS).
* Economic evaluation / cost-effectiveness (iPCQ).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a craniotomy.
2. Adult patients (cq age ≥18 years)
3. Sufficient knowledge of the Dutch language to understand the study documents in the judgement of the attending physician or researcher.
4. Provision of written informed consent by patient or legal representative.

Exclusion Criteria:

1. Impaired awareness before surgery (i.e. GCS < M6).
2. Planned post-operative ICU admission.
3. Suspected delirium (defined as fluctuating awareness).
4. Current antipsychotic treatment
5. Patients undergoing interventions impeding supply of music (e.g. surgical translabyrinthine approach, awake surgery).
6. Severe bilateral hearing impairment, defined as no verbal communication possible.
7. Current participation in other clinical trials interfering with results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-07-09 (Estimated); Study Completion 2023-03-09 (Estimated)

PRIMARY OUTCOMES:
Delirium | First five post-operative days. In case of discharge within 5 days towards home without delirium, it will be considered as no delirium.
  All participating patients on the ward will be screened using the Delirium Observation Screening (DOS) scale. The DOS is a score of 1 until 13, in which a score of 3 or higher is suspicious for delirium. Screening is conducted 3 times per day (i.e. during each shift) and maintained until day 5. In case of raised suspicion of delirium by DOS, a psychiatrist is consulted to confirm or reject clinical diagnosis of delirium based on the DSM-V criteria. Presence of delirium is confirmed by the psychiatrist after positive DOS screening, all other patients will be considered as absence of delirium. In case of discharge towards another hospital within 5 days, onset of delirium is evaluated in that hospital. In case of discharge within 5 days towards home without delirium, it will be considered as no delirium.

SECONDARY OUTCOMES:
Severity and duration of delirium. | First five days or discharge. In case of positive delirium until it has 'faded out'.
  In case of positive delirium, its severity will be assessed using the Delirium Rating Scale-revised-98 (DRS-R-98). DSR-98 regards a 13-item score sheet in which 0 represents the lowest and 39 represents the highest severity. It will be assessed by the consultant psychiatrist on the day of onset of delirium. Subsequently, as long as the delirium lasts the severity is assessed once every three days (i.e. Monday, Wednesday and Friday). To assess duration of delirium, the DOS score will be used; a DOS <3 during 24 hours will be considered as a 'faded out' delirium and number of days from onset until end will be documented.

OTHER OUTCOMES:
Pre-operative anxiety. | Day before surgery only
  Using the VAS-anxiety scale, a 11-numeric scale in which 0 represents no anxiety and 10 represents the worse imaginable anxiety, which is easy to use and highly correlated with the State-Trait Anxiety Inventory (STAI).
Activation of the parasympathetic nervous system. | The day of surgery (day 0) before and after surgery
  Heart rate variability (HRV), the variation in the time interval between adjacent heartbeats, with ECG recordings.
Depth of anesthesia with Bispectral Index. | During surgery
  Bispectral Index (BIS) which signal reflects processed brain activity, monitored by EEG and generated into numerical values. The acquired BIS value, ranging from 0 to 100, during anaesthesia provides information about the depth of anaesthesia. BIS-values are not evaluated during surgery but merely used for research purposes.
Peri-operative medication. | During admission.
  Peri-operative medication use, such as opioids, benzodiazepines and antipsychotic drugs will be extracted from the electronic patient files. Analgesic opioid medica-tion will be converted to milligrams of morphine equivalents, using a conversion tool based on the guidelines by the American Pain Society.61
Postoperative pain. | Post-operative day 1 - 3
  Postoperative pain, assessed using an 11-point NRS-scale, in which 0 implies no pain and 10 the worst pain possible.
Patients with postoperative complications. | Within two weeks after surgery.
  Postoperative complications such as post-operative hemorrhagic, surgical site infection, hydrocephalus, vasospasms, liquor leakage, epilepsy, pulmonary complications, thromboembolic complications, gastro-intestinal complications and urinary tract infections will be extracted from the electronic patient files. Definition of the complication is an adverse event within two weeks after surgery resulting in prolongation of current admission, new treatment (surgery or pharmacological) or death.
Hospital length of stay. | From baseline until discharge in the same admission having received the intervention.
  Peri-operative length of in-hospital stay in days.
Cognitive function. | Baseline, 3 months and 6 months after surgery.
  Cognitive function assessed with the Montreal Cognitive Assessment (MoCA) tool at baseline and during follow-up at 3 and 6 months. The MoCA is a validated 0 to 30 points scoring system involving visuospatial, naming, memory, language, abstraction, delayed recall and orientation.
Patient functional outcome. | Baseline, 6 weeks, 3 months and 6 months.
  Patient functional outcome expressed in Karnofsky Performance Scale (KPS). The KPS has achieved the reputation of 'gold standard' for the measurement of physical performance in clinical (neuro-) oncology. It consists of 11 categories denoted in deciles from 100 (asymptomatic, normal function) to 0 (death).
Patient functional outcome. | Baseline, 6 weeks, 3 months and 6 months.
  Patient functional outcome expressed in Modified Ranking Scale (mRS). The mRS is a 7-item scale from 0 (no symptoms) to 6 (dead) and is validated in patient groups with neurological diseases.
Mortality and readmission rate. | Follow up until 6 months.
  Mortality and readmission rate will be evaluated during the follow-up at 6 weeks, 3 and 6 months.
Patient reported outcome. | Baseline, 6 weeks, 3 months and 6 months after surgery.
  Patient reported outcomes, measured through the questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Cancer (EORTC QLQ-C30). The EORTC QLQ-C30, an approach for evaluating the Health-related quality of life (HRQoL) in international cancer clinical trials, incorporates nine multi-item scales: five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties). Items are presented as questions on a scale ranging from 1 = "not at all" to 4 = "very much."
Patient reported outcome. | Baseline, 6 weeks, 3 months and 6 months after surgery.
  Patient reported outcomes, measured through the questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Brain Neoplasm (EORTC BN-20). The EORTC BN-20, an approach for evaluating the Health-related quality of life (HRQoL) in patients with brain tumours, consists of 20 items that assess future uncertainty, visual disorder, motor dysfunction, and communication deficit. Items are presented as questions on a scale ranging from 1 = "not at all" to 4 = "very much."
Patient reported outcome. | Baseline, 6 weeks, 3 months and 6 months after surgery.
  Patient reported outcomes, measured through the EuroQol-5D (EQ-5D) questionnaire. The EQ-5D-3L, an approach for evaluating the Health-related quality of life (HRQoL) in patients, comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, moderate problems and extreme problems
Patient satisfaction. | Follow-up 6 weeks
  Patient satisfaction of music around operations will be measured through a Visual Analogue Scale: a line of 10 centimeters in length with "not satisfied at all" and "very satisfied" at the left and right extremes respectively.
Economic evaluation. | Follow-up at 3 and 6 months
  Productivity losses will be measured and valued using the iMTA Productivity Cost Questionnaire (iPCQ) collected at 3 and 6 months. The iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work.

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Dirven TLA, Kappen PR, van der Beek FTH, van der Holt B, Jeekel H, Dirven CMF, Vincent AJPE, Klimek M, Poley MJ. The effect of music interventions compared to standard-of-care on the prevention of delirium in neurosurgical patients: an analysis of costs and cost-effectiveness based on the MUSYC-trial. Acta Neurochir (Wien). 2025 Feb 14;167(1):46. doi: 10.1007/s00701-025-06448-0. PMID 39951210
- [Derived] Kappen PR, Mos MI, Jeekel J, Dirven CMF, Kushner SA, Osse RJ, Coesmans M, Poley MJ, van Schie MS, van der Holt B, Klimek M, Vincent AJPE. Music to prevent deliriUm during neuroSurgerY (MUSYC): a single-centre, prospective randomised controlled trial. BMJ Open. 2023 Jun 27;13(6):e069957. doi: 10.1136/bmjopen-2022-069957. PMID 37369412
- [Derived] Kappen P, Jeekel J, Dirven CMF, Klimek M, Kushner SA, Osse RJ, Coesmans M, Poley MJ, Vincent AJPE. Music to prevent deliriUm during neuroSurgerY (MUSYC) Clinical trial: a study protocol for a randomised controlled trial. BMJ Open. 2021 Oct 1;11(10):e048270. doi: 10.1136/bmjopen-2020-048270. PMID 34598983